CLINICAL TRIAL: NCT00865865
Title: Computer Aided Gap Balancing Improves Sagittal Stability and Outcomes for Cruciate-Retaining Total Knee Arthroplasty- 2-Year Results of a Prospective Randomised Trial
Brief Title: Computer Aided Gap Balancing Improves Sagittal Stability and Outcomes for Cruciate-Retaining Total Knee Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Responsible Party: DR SENG-JIN YEO, Singapore General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: #48/2006
Record Dates: First submitted 2009-03-17; First posted 2009-03-19 (Estimated); Last update posted 2009-03-19 (Estimated); Status verified 2009-03

CONDITIONS: Osteoarthritis of the Knee
Keywords: Knee; Computer; Gap; Soft tissue; Balancing; Replacement; Arthroplasty
MeSH Terms: conditions — Osteoarthritis, Knee; Capillary Malformation-Arteriovenous Malformation | interventions — Surgery, Computer-Assisted

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Other): Conventional total knee arthroplasty
  Interventions: Procedure: Conventional total knee arthroplasty
- 2 (Active Comparator): Computer aided total knee arthroplasty
  Interventions: Procedure: Computer aided total knee arthroplasty

INTERVENTIONS:
Procedure: Computer aided total knee arthroplasty — Use of computer aided surgery to balance soft tissue tension in total knee arthroplasty
  Other Names: Computer aided surgery
  Arms: 2
Procedure: Conventional total knee arthroplasty — Conventional method of total knee arthroplasty
  Arms: 1

SUMMARY:
Computer Aided Surgery in total knee arthroplasty improves knee stability and functional outcomes more than conventional total knee arthroplasty.

DETAILED DESCRIPTION:
The success of total knee arthroplasty depends on restoration of limb alignment, precise implant positioning and optimal gap balancing. The advent of computer aided surgery (CAS) has improved limb alignment and implant positioning. The objective of this study was to evaluate the functional outcome of computer aided soft tissue gap balancing in total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria:

* primary osteoarthritis of the knee

Exclusion Criteria:

* rheumatoid arthritis, previous knee surgery, infection and those who could not be treated with unconstrained cruciate retaining TKA and a short stem tibial implant

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2006-05; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Sagittal stability of knee | 2 YEARS

SECONDARY OUTCOMES:
Functional status of postoperative patients | 2 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: SENG-JIN YEO, FRCS, Principal Investigator — Singapore General Hospital